CLINICAL TRIAL: NCT06811441
Title: Third Wave of the EVAL-PLH (POLYhandicap) Cohort: New Eyes
Acronym: EVAL-POLYNE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23_0252
Record Dates: First submitted 2025-01-30; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Polyhandicap

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general objective of the EVAL-PolyNE project is to improve the representativeness of the EVAL-PLH cohort by broadening participation in the John Bost Foundation, due to its geographical particularity and its private valence.

DETAILED DESCRIPTION:
Studies on people with profound intellectual and multiple disabilities (PIMD)/Polyhandicap are rare, involve small numbers and highly heterogeneous groups, and document narrow objectives focused on targeted health problems. Although valuable, these studies provide only fragmentary knowledge of the medical, socio-economic and epidemiological determinants of the health and experience of people with PIMD/Polyhandicap and their families. Existing studies are based on retrospective or cross-sectional data. These study designs do not make it possible to identify causal links between the phenomena observed. Only cohort studies can provide a longitudinal vision, enabling us to study the dynamics of the phenomena observed (care, access to different care structures, environment in the broadest sense, state of health and experiences of these people and their families). The information made available is essential for informing healthcare decision-makers, healthcare professionals and the families of these people, and for proposing the most appropriate targeted actions.

The Eval-PLH cohort of people with PIMD/Polyhandicap was initiated in 2015, with the aim of describing prospective changes in the health characteristics of people with PIMD/Polyhandicap, clinical practices and management strategies for PIMD/Polyhandicap. It also assesses the impact of PIMD/Polyhandicap on the experiences of family carers and the institutional carers (caregivers) who support them.

The 1st wave of observation took place in 2015-2016. Nearly 900 people with PIMD/Polyhandicap, 400 family carers and 400 institutional carers were assessed thanks to the participation of six specialized follow-up care and rehabilitation centers, eight medico-social structures (MAS and IME) and one neuropediatric consultation service. Data mining has enabled us to build up an unprecedented knowledge base. This work confirmed the diversity and evolution of pathologies, the heterogeneity of medical practices and the impact on family and institutional caregivers.

The 2nd wave of observation took place in 2020-2021 and assessed 624 people PIMD/Polyhandicap (132 new cases, 492 cases present in the 1st wave), 226 family carers and 223 institutional carers in four specialized follow-up care and rehabilitation centers and eight medico-social structures. These data are currently being explored and valorized. They provide considerable scientific added value thanks to their longitudinal perspective. A more detailed understanding of the phenomena (through a qualitative approach based on interviews) complements the initial purely quantitative approach.

The present study, which concerns the 3rd evaluation wave, aims to optimize the system, particularly in terms of the representativeness of the populations studied. The extension of the system to less targeted geographical areas and to non-public structures will shed new light on the care organizations and professionals affiliated with these structures, as well as on the experiences of the people cared for (patients and families).

ELIGIBILITY:
Inclusion Criteria:

* Patient with PIMD/Polyhandicap
* Patient for whom the legal representative has received the information note of the EVAL-PLH cohort and has not expressed opposition to the collection of patient data;
* Patient aged at least 3 years;
* Patient affiliated to a health insurance scheme;
* Patient treated within the department of the participating center;
* Patient for whom the legal representative understands the French language;
* Patient with a PIMD/Polyhandicap

Family caregivers of patient

* Subject identified by the care structure as the reference family caregiver;
* Subject aged at least 18 years;
* Subject who understands the French language and is able to complete self-questionnaires;
* Subject who has received the information notice and has not expressed opposition to participating in this project

Institutinal caregivers of patient

* Subject identified by the care structure as the reference institutional caregiver of at least one patient included in this project;
* Subject aged at least 18 years;
* Subject who understands the French language and is able to complete self-questionnaires;
* Subject who has received the information notice and has not expressed opposition to participating in this project.

Exclusion Criteria:

* Patient with PIMD/Polyhandicap
* Patient not meeting all inclusion criteria;
* Patient in exclusion period of another research protocol at the time of inclusion.

Family and Institutional caregivers of patient

• Subject not meeting all inclusion criteria

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a PIMD/Polyhandicap defined according to the following criteria:
  * Presence of a brain lesion that occurred before the age of 3,
  * IQ below 40 or not assessable,
  * Motor handicap: para/tetraparesis or hemiparesis,
  * Gross Motor Function Classification System score of III, IV or V,
  * Functional Independence Measure score below 55
Sampling Method: Non-Probability Sample
Enrollment: 1102 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Health status of patients with PIMD/Polyhandicap | 2 hours to complete the questionnaire
  Evaluate the health status of patients with PIMD/Polyhandicap using a standardized questionnaire completed by a physician.

SECONDARY OUTCOMES:
Quality of life of patients with PIMD/Polyhandicap | 10 minutes to complete the questionnaire
  Evaluate the quality of life of patients with PIMD/Polyhandicap using a standardized questionnaire completed by institutional caregivers and family caregivers
Health status and quality of life of family caregivers | 1 hour to complete the self-reported questionnaire
  Evaluate the health status and quality of life of family caregivers using a standardized self-reported questionnaire
Health status and quality of life of institutional caregivers | 30 minutes to complete the self-reported questionnaire
  Evaluate the health status and quality of life of institutional caregivers using a standardized self-reported questionnaire
Evolution of the health status of patients, clinical practices and management strategies | 2 hours to complete the patient questionnaire by the physician / 1 hour to complete the family caregiver self-reported questionnaire / 30 minutes to complete the institutional caregiver self-reported questionnair
  Identify the determinants of health status and quality of life of patients with PIMD/Polyhandicap, family and institutional caregivers using standardized questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: karine Baumstarck, Principal Investigator — Assistance Publique des Hôpitaux de Marseille (AP-HM)
Locations (6):
- France (6):
  - Hôpital Marin de Hendaye, Hendaye
  - Hôpital San Salvadour, Hyères
  - Fondation John Bost, La Force
  - Assistance Publique Des Hopitaux de Marseille, Marseille
  - CESAP, Paris
  - Hôpital La Roche Guyon, Paris